CLINICAL TRIAL: NCT01950039
Title: Bedside to Bench and Back: Cardiometabolic Effects of Betaine Supplementation
Brief Title: Metabolic Effects of Betaine Supplementation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2013P001265; 7-13-CE-17 (Other Grant/Funding Number: American Diabetes Association 7-13-CE-17)
Record Dates: First submitted 2013-09-16; First posted 2013-09-25 (Estimated); Results first posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-03

CONDITIONS: Obesity; Dysglycemia
Keywords: Obesity; Glucose Intolerance
MeSH Terms: conditions — Obesity; Glucose Intolerance | interventions — Betaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Betaine (Active Comparator)
  Interventions: Drug: Betaine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Betaine — Betaine or placebo administered orally in divided doses over 12 weeks
  Other Names: trimethyl glycine
  Arms: Betaine
Drug: Placebo — Placebo administered orally in divided doses over 3 months
  Arms: Placebo

SUMMARY:
Betaine is important in cellular metabolic pathways. Few epidemiologic studies link betaine levels to diabetes and cardiovascular disease. Small human studies suggest benefit for non-alcoholic liver disease. In this study we will determine if administration of betaine improves metabolic measures, liver fat and/or endothelial function in humans with glucose intolerance who are overweight.

DETAILED DESCRIPTION:
This study is a single site, prospective, randomized (1:1), double masked, placebo controlled trial to assess metabolic effects of betaine compared to placebo on glycemia and insulin sensitivity, liver fat and endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* 1) Men and women aged 21-65 years old;
* 2) Dysglycemia/prediabetes is defined as impaired fasting glucose (≥100 mg/dl), impaired glucose tolerance (2 hour post 75 g oral glucose load 140-200 mg/dl) or HbA1c 5.7-6.5%);
* 3) overweight to grade 3 obesity (BMI 25 to 45 kg/m2).

Exclusion Criteria:

* 1) cystathionine beta-synthase (CBS deficiency);
* 2) Presence of liver disease other than NAFLD;
* 3) Use of medications causing steatosis;
* 4) Known alcohol consumption ≥ 2 drink per day;
* 5) Use of medications known to cause insulin resistance;
* 6) Use of weight loss drugs (or program) within 3 months of screening;
* 7) Treatment with any experimental drug within the past 6 months;
* 8) Subjects must be willing to abstain from use of phosphodiesterase type 5 (PDE-5) inhibitors;
* 9) Pregnancy or lactation, and women of child bearing potential must use adequate contraception;
* 10) Surgery within 30 days of screening;
* 11) Heart disease defined as New York Heart Association Class III or IV cardiac status or hospitalization for congestive heart failure, unstable angina, myocardial infarction, cerebrovascular accident, transient ischemic attack or any revascularization within 6 months;
* 12) Uncontrolled hypertension;
* 13) eGFR <60; 14) History of acquired immune deficiency syndrome;
* 15) History of malignancy within 5 years;
* 16) Hemoglobin <12 g/dL (males), <10 g/dL (females);
* 17) Triglycerides (TG) >500 mg/dL;
* 18) Poor mental function or any other reason to expect patient difficulty in complying with study requirements;
* 19) Metal clips or implants that preclude magnetic resonance imaging.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Joslin Diabetes Center and Brigham and Womens Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Grizales AM, Patti ME, Lin AP, Beckman JA, Sahni VA, Cloutier E, Fowler KM, Dreyfuss JM, Pan H, Kozuka C, Lee A, Basu R, Pober DM, Gerszten RE, Goldfine AB. Metabolic Effects of Betaine: A Randomized Clinical Trial of Betaine Supplementation in Prediabetes. J Clin Endocrinol Metab. 2018 Aug 1;103(8):3038-3049. doi: 10.1210/jc.2018-00507. PMID 29860335

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study subjects with overweight and T2D risk factors were screened for dysglycemia and enrolled at 1 site in the US.
Groups:
- Betaine: Betaine:
  Participants were instructed to take betaine 3300 mg (10 ml) orally twice daily for 10 days, then 4950 mg (15 ml) orally twice daily through 12 weeks.
- Placebo: Placebo: Participants were instructed to take identical amounts and appearance of placebo through 12 weeks.
Period: Overall Study
Arm/Group | Betaine | Placebo
Started | 15 | 13
Study Drug Initiated | 14 | 13
Completed Clamp | 13 | 12
Completed MRI | 13 | 12
Completed Endothelial Evaluation | 14 | 12
Completed | 14 | 13
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline clinical characteristics were similar between groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Betaine | Placebo | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (7) | 57 (8) | 59 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 10 | 9 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and Ethnicity: Asian | 2 | 0 | 2
  Race and Ethnicity: Black or African American | 3 | 2 | 5
  Race and Ethnicity: White | 7 | 11 | 18
  Race and Ethnicity: Hispanic | 2 | 0 | 2
Region of Enrollment [Number; unit: participants] — Participants were recruited from the New England region.
  participants
    United States | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Fasting and 2 Hour Glucose Levels, Comparing Baseline and 12 Weeks.
Description: Glucose levels were analyzed in the fasting state and two hours after glucose load, comparing baseline to 12 weeks.
Time Frame: baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Betaine | Placebo
Number analyzed (Participants) | 14 | 13
mg/dl
  fasting glucose | -5 [-12 to 1] | 3 [-4 to 9]
  2-hour glucose | 7 [-10 to 25] | -4 [-22 to 13]

2. Primary Outcome: Change in Glucose AUC at 12 Weeks From Baseline (Glucose Tolerance)
Description: Glucose tolerance was assessed by oral glucose tolerance, assessed using the change from baseline for fasting and 2 hour glucose, and change in Glucose AUC at 12 weeks from baseline was measured.
Time Frame: baseline and 12 weeks
Measure: Mean (95% Confidence Interval); unit: mg*min/dL
Arm/Group | Betaine | Placebo
Number analyzed (Participants) | 14 | 13
mg*min/dL | 340 [-993 to 1672] | -413 [-1749 to 923]

3. Primary Outcome: Hepatic Fat, Change From Baseline
Description: Intrahepatic triglyceride levels were assessed by magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (Siemens 3T TIM Skyra, software version VD13; Siemens, Erlangen, Germany).
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Error); unit: percent change in hepatic triglyceride
Arm/Group | Betaine | Placebo
Number analyzed (Participants) | 13 | 12
percent change in hepatic triglyceride | -0.01 (0.02) | -0.03 (0.02)

4. Primary Outcome: Endothelial Function
Description: Brachial artery reactivity to flow and nitroglycerin stimuli, assessed as percent change from baseline
Time Frame: baseline and 12 weeks
Population: One participant in the placebo group was not able to complete nitroglycerine-mediated dilation assessment.
Measure: Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Betaine | Placebo
Number analyzed (Participants) | 14 | 13
percent change from baseline
  Percent change in flow-mediated dilation | -0.5 [-3.3 to 2.3] | -1.9 [-4.7 to 1.0]
  Percent change in nitroglycerine-mediated dilation: number analyzed (Participants) | 14 | 12
  Percent change in nitroglycerine-mediated dilation | -0.9 [-4.0 to 2.1] | -0.9 [-4.1 to 2.4]

5. Primary Outcome: Insulin Sensitivity
Description: Euglycemic hyperinsulinemic clamp at baseline and at end of study (12 weeks) for assessment of:
  1. glucose disposal (M) at low (25 mU/m2/min) and high (180 mU/m2/min) insulin infusion rates, reported as raw data
  2. measurement of endogenous glucose production at basal and low insulin infusion (25 mU/m2/min), reported as change from measures at baseline of individual study days
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: umol/kg/min
Arm/Group | Betaine | Placebo
Number analyzed (Participants) | 13 | 12
umol/kg/min
  Glucose Utilization (M), 25 mU/m2/min, baseline | 90.4 (16.5) | 62.8 (13.5)
  Glucose Utilization (M), 25 mU/m2/min, 12 weeks | 110.9 (16.9) | 73.5 (13.8)
  Glucose Utilization (M), 180 mU/m2/min, baseline | 406.8 (30.4) | 332.6 (39.1)
  Glucose Utilization (M), 180 mU/m2/min, 12 weeks | 458.1 (38.7) | 393.7 (44.1)
  Endogenous Glucose Production, basal insulin | .03 (.09) | -0.01 (0.09)
  Endogenous Glucose Production, 25 mU/m2/min | -0.01 (0.12) | -0.12 (0.13)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 14 weeks (during study drug administration and for 2 weeks after last study drug).
Arm/Group | Betaine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 4/14 | 6/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Betaine (N=14) | Placebo (N=13)
Irritation (Eye disorders) | 0 (0) | 1 (1)
GI infection (Gastrointestinal disorders) | 0 (0) | 1 (1)
GI motility and defecation conditions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatic and hepatobiliary disorders (Hepatobiliary disorders) | 1 (1) | 0 (0)
Immune disorders (Immune system disorders) | 0 (0) | 1 (1)
Metabolism and nutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract signs and symptoms (Renal and urinary disorders) | 0 (0) | 1 (2)
Respiratory disorders NEC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract infections (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-09-19): https://cdn.clinicaltrials.gov/large-docs/39/NCT01950039/Prot_000.pdf
  • Statistical Analysis Plan (2014-01-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT01950039/SAP_001.pdf